CLINICAL TRIAL: NCT00004037
Title: Evaluation of Docetaxel in Recurrent, Platinum Resistant, Refractory and Paclitaxel Refractory Ovarian Cancer and Primary Peritoneal Carcinoma
Brief Title: Docetaxel in Treating Patients With Recurrent or Refractory Ovarian or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066369; GOG-126J
Record Dates: First submitted 1999-12-10; First posted 2003-06-25 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2003-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel in treating patients with recurrent or refractory ovarian or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the antitumor activity of docetaxel in patients with paclitaxel- and platinum-resistant, recurrent or refractory, ovarian epithelial or primary peritoneal cancer who have failed on higher priority treatment protocols. II. Determine the nature and degree of toxicity of docetaxel in this patient population.

OUTLINE: Patients receive docetaxel as a 1 hour continuous intravenous infusion. Courses are repeated every 21 days. Treatment continues in the absence of unacceptable toxic effects or disease progression. All patients are followed every 3 months for 2 years, every 6 months for 3 years, and then until death.

PROJECTED ACCRUAL: A total of 23-56 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or refractory ovarian epithelial or peritoneal cancer Platinum resistant AND paclitaxel resistant Progressed on or within 6 months of completing therapy with paclitaxel and platinum either alone or in combination Bidimensionally measurable disease (excludes ascites and pleural effusions) Brain metastases allowed provided that other measurable disease exists and brain lesions required no therapy for 6 months and are not life threatening Not eligible for higher priority GOG protocol

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT/SGPT no greater than 1.5 times ULN Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: No significant infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of allergic reaction to polysorbate 80 (e.g., etoposide or vitamin E) No other invasive malignancies within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Must have had at least 1 prior platinum based chemotherapeutic regimen containing carboplatin, cisplatin, or another organoplatinum compound Must have had at least 1 prior paclitaxel based chemotherapeutic regimen 1 or 2 prior chemotherapy regimens containing platinum and paclitaxel allowed Recovered from toxic effects No prior docetaxel Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Recovered from effects of recent surgery Other: At least 3 weeks since any prior therapy directed at the malignant tumor No prior cancer treatment that contraindicates this protocol therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Study Chair — The Cleveland Clinic
Locations (67):
- United States (66):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brookview Research, Inc., Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada

REFERENCES:
- [Result] Rose PG, Blessing JA, Ball HG, Hoffman J, Warshal D, DeGeest K, Moore DH. A phase II study of docetaxel in paclitaxel-resistant ovarian and peritoneal carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2003 Feb;88(2):130-5. doi: 10.1016/s0090-8258(02)00091-4. PMID 12586591